CLINICAL TRIAL: NCT04282824
Title: Evaluation by 68Ga-PSMA-11 PET Imaging of Monosodium Glutamate as a Potential Agent for Salivary Gland Protection Under PSMA-targeted Alpha-therapy: a Randomized Pilot Imaging Research Study
Brief Title: Impact of Monosodium Glutamate on 68GA-PSMA-11, PET Imaging Biodistribution in Patients With Prostate Cancer
Acronym: MSG PSMA PET
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18-001776; NCI-2019-04437 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-001776 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Sodium Glutamate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (68GA-PSMA-11, PET/CT, monosodium glutamate) (Experimental): 8 patients receive gallium Ga 68-labeled PSMA-11 IV and PET/CT scan on day 1. Within 2 weeks (days 2-14), patients receive MSG PO over 10 minutes and receive a second dose of gallium Ga 68-labeled PSMA-11 IV, followed by a second PET/CT scan. Patients also undergo collection of saliva at 0, 30, and 60 minutes after gallium Ga 68-labeled PSMA-11 injection and 90 minutes after PET/CT.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Gallium Ga 68-labeled PSMA-11; Dietary Supplement: Monosodium Glutamate; Procedure: Positron Emission Tomography
- Arm II (68GA-PSMA-11, PET/CT, monosodium glutamate) (Experimental): 8 patients receive gallium Ga 68-labeled PSMA-11 IV and undergo a PET/CT scan on day 1. Within 2 weeks (days 2-14), patients receive a second dose of gallium Ga 68-labeled PSMA-11 IV immediately followed by MSG applied in the mouth over 30 seconds every 10 minutes for a total of 6 times, and then undergo a second PET/CT scan. Patients also undergo collection of saliva at 0, 30, and 60 minutes after gallium Ga 68-labeled PSMA-11 injection and 90 minutes after PET/CT.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Gallium Ga 68-labeled PSMA-11; Dietary Supplement: Monosodium Glutamate; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of saliva
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT scan; tomography
Drug: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Dietary Supplement: Monosodium Glutamate — Given PO
  Other Names: MSG Monohydrate; Sodium Glutamate Monohydrate
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies the impact of monosodium glutamate (MSG) on 68GA-PSMA-11 PET/CT in decreasing the salivary glands uptake in patients with prostate cancer. Prostate specific membrane antigen (PSMA) is a molecule that is overexpressed by the prostate cancer cells. 68GA-PSMA-11 is an imaging radioactive drug that can target this molecule in tissues for imaging and therapy of prostate cancer. Food substances, such as monosodium glutamate, may reduce salivary gland uptake of 68GA-PSMA-11. Ultimately, giving MSG may reduce potential harm and injury to the salivary glands in patients with prostate cancer treated with PSMA-targeted molecular radiotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of monosodium glutamate (MSG) administration (glutamate supplementation) on the salivary gland uptake of gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11).

SECONDARY OBJECTIVES:

I. To determine the effect of MSG administration on renal 68Ga-PSMA-11 uptake. II. To determine the effect of MSG administration on tumor 68Ga-PSMA-11 uptake. III. To determine if 68GA-PSMA-11 is excreted in the saliva. IV. Safety of MSG administration both oral ingestion and oral-salivary stimulation.

OUTLINE: Patients are randomized to 1 of 2 arms.

Arm I: Patients receive gallium Ga 68-labeled PSMA-11 intravenously (IV) and undergo a positron emission tomography (PET)/computed tomography (CT) scan on day 1. Within 2 weeks (days 2-14), patients receive MSG orally (PO) over 10 minutes and receive a second dose of gallium Ga 68-labeled PSMA-11 IV, followed by a second PET/CT scan. Patients also undergo collection of saliva at 0, 30, and 60 minutes after gallium Ga 68-labeled PSMA-11 injection and 90 minutes after PET/CT.

Arm II: Patients receive gallium Ga 68-labeled PSMA-11 IV and undergo a PET/CT scan on day 1. Within 2 weeks (days 2-14), patients receive a second dose of gallium Ga 68-labeled PSMA-11 IV immediately followed by MSG applied in the mouth over 30 seconds every 10 minutes for a total of 6 times, and then undergo a second PET/CT scan. Patients also undergo collection of saliva at 0, 30, and 60 minutes after gallium Ga 68-labeled PSMA-11 injection and 90 minutes after PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Patient volunteer to undergo 2 PSMA PET/CT scans within 14 days
* Histopathologically proven prostate cancer (PCa)
* PSMA PET/CT indicated for :

  * Initial staging before definitive therapy
  * Biochemical recurrence localization
  * Metastatic disease re-staging
* Ability to understand a written informed consent document and the willingness to sign it
* Ability to ingest 300 mL of fluid across 10 minute period

Exclusion Criteria:

* Prior salivary gland surgery or radiation therapy
* Prior history or current salivary gland disease
* Unable to lie flat, still or tolerate a PET scan
* Unable to follow the salivary flow stimuli administration regimen
* Unable to follow the glutamate supplementation administration regimens
* Asthma
* Severe uncontrolled hypertension (systolic blood pressure above 140 mm Hg and diastolic blood pressure above 90 mm Hg, or systolic blood pressure above 180 mm Hg, or diastolic blood pressure above 110 mg Hg). Patients with controlled hypertension under medication are eligible
* Sodium/salt restricted diet due to other medical conditions
* History of severe asthma that has led to hospitalizations or emergency room visits
* History of severe contraindications to MSG consumption including severe headaches, migraines or other intolerance
* Change to treatment administered between time of baseline scan and MSG scan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Salivary gland uptake of gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) | 2 measurements within 2 to 14 days maximum (on positron emission tomography [PET]1 and PET2)
  Standard uptakes values (SUV) values (maximum SUV [SUVmax] and SUVmean) in all assessable salivary glands will be measured with a spherical volume-of-interest with and without the administration of monosodium glutamate (MSG) interventions. SUVmax/salivary gland will be calculated and a mean SUVmax/patient will be generated. The aim is to show a 2-fold reduction of the salivary gland 68Ga-PSMA-11 uptake after MSG administration. Paired T-test will be used to determine statistical significance per salivary gland and per patient.

SECONDARY OUTCOMES:
Renal 68Ga-PSMA-11 uptake | 2 measurements within 2 to 14 days maximum (on PET1 and PET2)
  SUVmax and SUVmean in the kidneys will be measured with a spherical volume-of-interest with and without the administration of MSG interventions. SUVmax/kidneys will be calculated and a mean SUVmax/patient will be generated. Paired T-test will be used to determine statistical significance per salivary gland and per patient.
Tumor 68Ga-PSMA-11 uptake | 2 measurements within 2 to 14 days maximum (on PET1 and PET2)
  SUVmax and SUVmean in the visible tumor lesions will be measured with a spherical volume-of-interest with and without the administration of MSG interventions. SUVmax/tumor lesions will be calculated and a mean SUVmax/patient will be generated. Paired T-test will be used to determine statistical significance per salivary gland and per patient.
Saliva radioactivity concentration | 2 measurements within 2 to 14 days maximum (on PET1 and PET2)
  Saliva radioactivity concentration will be compared with and without saliva stimuli.
Incidence of adverse events of MSG administration | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, M.D., Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States